CLINICAL TRIAL: NCT00004442
Title: Study of Bile Acids in Patients With Peroxisomal Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13442; CHMC-C-FDR000995
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-11

CONDITIONS: Infantile Refsum's Disease; Zellweger Syndrome; Bifunctional Enzyme Deficiency; Adrenoleukodystrophy
Keywords: Zellweger syndrome; adrenoleukodystrophy; bifunctional enzyme deficiency; inborn errors of metabolism; infantile Refsum's disease; peroxisomal disorders; pseudo-Zellweger syndrome; rare disease; sphingolipidoses
MeSH Terms: conditions — Refsum Disease, Infantile; Zellweger Syndrome; Pseudo-Zellweger syndrome; Adrenoleukodystrophy; Metabolism, Inborn Errors; Peroxisomal Disorders; Rare Diseases; Sphingolipidoses | interventions — Chenodeoxycholic Acid; Cholic Acid; Ursodeoxycholic Acid

INTERVENTIONS:
Drug: chenodeoxycholic acid
Drug: cholic acid
Drug: ursodiol

SUMMARY:
OBJECTIVES: I. Determine the effectiveness of oral bile acid therapy with cholic acid, chenodeoxycholic acid, and ursodeoxycholic acid in patients with peroxisomal disorders involving impaired primary bile acid synthesis.

II. Determine whether suppression of synthesis of atypical bile acids and enrichment of bile acid pool with this regimen is effective in treating this patient population and improving quality of life.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive oral cholic acid and oral chenodeoxycholic acid on day 1. On day 4, patients receive oral cholic and ursodeoxycholic acids. Patients are assessed at 3 and 6 months for liver function response, neurologic status, and nutritional status.

Patients receive treatment until disease progression or unacceptable toxic effects are observed.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Biochemically proven peroxisomal disorder, including:

* Zellweger syndrome
* Pseudo-Zellweger syndrome
* Neonatal adrenoleukodystrophy
* Bifunctional enzyme deficiency
* Infantile Refsum's disease

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Study Completion 1999-04

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Setchell, Study Chair — Children's Hospital Medical Center, Cincinnati